CLINICAL TRIAL: NCT02116699
Title: Oropharyngeal Administration of Mother's Colostrum: Health Outcomes of Premature Infants
Brief Title: Oropharyngeal Administration of Mother's Colostrum for Premature Infants (NS-72393-360)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: The Gerber Foundation (Other); Fundacion Para La Investigacion Hospital La Fe (Other); University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EH11-360
Record Dates: First submitted 2014-04-11; First posted 2014-04-17 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Infection; Enterocolitis, Necrotizing; Ventilator-associated Pneumonia
Keywords: oropharyngeal; colostrum; mother's milk; premature; neonate; infection; necrotizing enterocolitis; ventilator-associated pneumonia; breastmilk; human milk; late-onset sepsis; microbiome; antioxidant; enteral feeds
MeSH Terms: conditions — Infections; Enterocolitis, Necrotizing; Pneumonia, Ventilator-Associated; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oropharyngeal mother's milk (Experimental): 0.2 mL every 2 hours for 48 hours beginning within 96 hours post-birth, followed by 0.2 mL every 3 hours until 32 weeks post conceptional age
  Interventions: Other: oropharyngeal mother's milk
- oropharyngeal sterile water (Placebo Comparator): 0.2 mL every 2 hours for 48 hours beginning within 96 hours post-birth, followed by 0.2 mL every 3 hours until 32 weeks post conceptional age
  Interventions: Other: oropharyngeal sterile water

INTERVENTIONS:
Other: oropharyngeal mother's milk — Application of 0.2 mL of own mother's milk onto the infant's oral mucosa, for an initial treatment period of every 2 hours for 48 hours, followed by an extended treatment period of every 3 hours until 32 weeks corrected gestational age
  Arms: oropharyngeal mother's milk
Other: oropharyngeal sterile water — Application of 0.2 mL of sterile water onto the infant's oral mucosa, for an initial treatment period of every 2 hours for 48 hours, followed by an extended treatment period of every 3 hours until 32 weeks corrected gestational age
  Arms: oropharyngeal sterile water

SUMMARY:
Extremely premature (BW<1250g) infants are at high risk for morbidity and mortality. Own mother's colostrum (OMC) and milk (OMM) protect against neonatal morbidity and are rich in immune factors which may provide immunostimulatory effects when administered oropharyngeally to extremely premature infants during the first weeks of life. The investigators hypothesize that infants who receive oropharyngeal mother's colostrum and milk will have significantly lower rates of infection and improved health outcomes, compared to infants who receive a placebo.

DETAILED DESCRIPTION:
Extremely premature (BW<1250g) infants are at high risk for morbidity and mortality. Own mother's colostrum (OMC) and milk (OMM) protect against neonatal morbidity and are rich in immune factors which may provide immunostimulatory effects when administered oropharyngeally to extremely premature infants during the first weeks of life. This 5-year placebo-controlled, double-blind randomized controlled trial will evaluate the safety, efficacy and health outcomes of oropharyngeal administration of OMC/OMM in a sample of 622 (total patients enrolled) extremely premature infants with the following aims: Aim 1. To determine if oropharyngeal administration of OMC/OMM to extremely premature infants will reduce the risk of late-onset sepsis or death as the primary outcome, and necrotizing enterocolitis and ventilator-associated pneumonia as pre-planned secondary outcomes. Aim 2: To determine if extremely premature infants who receive OMC/OMM via the oropharyngeal route have a shorter time to reach full enteral feeds and a shorter length of hospital stay. Aim 3: To determine if oropharyngeal administration of OMC/OMM will have immunostimulatory effects for extremely premature infants, as measured by (A) enhancement of gastrointestinal (fecal) microbiota, (B) improvement in antioxidant defense maturation or reduction of pro-oxidant status, and (C) maturation of immunostimulatory effects as measured by changes in urinary lactoferrin. Results will confirm whether extremely premature infants demonstrate a host-immune response to this intervention and whether there is a beneficial effect on common morbidities in these high risk patients.

ELIGIBILITY:
Inclusion Criteria:

Birthweight <1250g Mother plans to pump and provide breastmilk for at least 2 months Absence of severe congenital anomalies Admission to the neonatal intensive care unit within 24 hours after birth Ability to begin protocol within 96 hours of life

Exclusion Criteria:

Gastrointestinal anomaly pH < 7.0 on initial blood gas in NICU Maternal +HIV status Maternal drug or substance use that precludes infant from receiving mother's milk Tracheoesophageal fistula

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2013-11-20 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Incidence of of late-onset sepsis | at 40 wks CGA
  positive blood cultures (not deemed contaminated) collected after 72 hours of age, and 2 clinical symptoms
Incidence of necrotizing enterocolitis | at 40 weeks CGA
  defined according to modified Bell's criteria stage >2 with clinical signs and radiological evidence of pneumatosis intestinalis or portal venous gas
Incidence of ventilator-associated pneumonia | at 40 weeks CGA

SECONDARY OUTCOMES:
Time to reach full enteral feeds | at 40 wks CGA
  defined as # days to reach a 120kcal/kg/day
Length of hospital stay | at 40 wks CGA
Concentrations of lactoferrin in urine | 1 day, 3 days, 32 weeks CGA
Changes in stool microbiome | 3 days, 2 weeks, 32 weeks CGA
Changes in urinary biomarkers of oxidative stress | 3 days,
  1 day, 3 days, 1 week, 32 weeks CGA

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Garofalo (previously Rodriguez), PhD APN NNP, Principal Investigator — Endeavor Health
Locations (5):
- United States (5):
  - South Miami Hospital, Miami, Florida
  - NorthShore University health System, Evanston, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Morristown Medical Center, Morristown, New Jersey
  - Betty Cameron Women & Children's Hospital, Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Rodriguez NA, Moya F, Ladino J, Zauk A, Prazad P, Perez J, Vento M, Claud E, Wang CH, Caplan MS. A randomized controlled trial of oropharyngeal therapy with mother's own milk for premature infants. J Perinatol. 2023 May;43(5):601-607. doi: 10.1038/s41372-022-01589-x. Epub 2023 Jan 3. PMID 36596945
- [Derived] Rodriguez NA, Vento M, Claud EC, Wang CE, Caplan MS. Oropharyngeal administration of mother's colostrum, health outcomes of premature infants: study protocol for a randomized controlled trial. Trials. 2015 Oct 12;16:453. doi: 10.1186/s13063-015-0969-6. PMID 26458907